CLINICAL TRIAL: NCT03519217
Title: Diabetes Mellitus Under the Age of One Year: Clinical Pattern, Etiological Factors and Possible Mutation in KCJN11 Gene Encoding of Adenosine Tri-phosphate Sensitive Potassium Channel Gene ( Kir6.2).
Brief Title: Genetic Study for Infantile Onset Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shimaa Kamal (Other)
Responsible Party: Sponsor-Investigator, Shimaa Kamal, Director, clinical research, Assiut University
Organization: Assiut University (Other)
Other Study IDs: INFANTILE DIABETES MELLITUS
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Gene Mutation in Infantile Onset Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Each patient with diabetes mellitus diagnosed under the age of one year( sixty patients) will be subjected to do Blood glucose level, glycated haemoglobin, fasting C- peptide, anti-insulin antibody, anti-islet antibody, and who have negative tests for anti-insulin and anti- islet will subjected to do genetic study for KCJN11 and ABCC8
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients under the age of one year: All cases which are diagnosed with diabetes mellitus under the age of one year will be subjected for blood glucose level, glycated haemoglobin, fasting C-peptide, anti-insulin and anti-islets auto-antibodies, and who have negative tests for anti-insulin and anti-islets auto-antibodies, will be subjected to do genetic study for KCJN11 and ABCC8

SUMMARY:
Diabetes mellitus is a group of metabolic diseases characterized by chronic hyperglycemia resulting from defects in insulin secretion, insulin action, or both.

DETAILED DESCRIPTION:
Infantile onset diabetes mellitus is not uncommon metabolic disorder in children, with rising in the incidence in the last few years. Infants with onset of diabetes mellitus at age less than one year are likely to have transient or permanent neonatal diabetes mellitus or rarely type one diabetes, all infants with onset of diabetes at less than one year of age need to undergo genetic evaluation for monogenic diabetes as is most commonly due to activating mutations in either of the genes encoding the two subunits of the adenosine tri-phosphate-sensitive potassium channel (potassium channel, inwardly rectifying subfamily J member 11 and adenosine tri-phosphate-binding cassette, sub-family C, member 8) as those patients will respond to therapy with sulphonylurea lead to good glycemic control and management of other comorbid factors. Evaluation with auto-immune antibodies may be warranted in infants with onset of diabetes in late infancy as the chances of type 1 diabetes presenting in late infancy has been reported in the literature.

Type 1 diabetes mellitus is one of the most common endocrine and metabolic conditions in childhood.

Data from large epidemiological studies worldwide indicate that on an annual basis, the overall increase in the incidence of type one diabetes is around three percent.

There is increase in incidence of type one diabetes mellitus throughout the world especially, marked in young children, Registries in Europe suggest that incidence of type one diabetes mellitus were highest in the youngest age-group (0-4 years).

The underlying pathophysiological mechanism of the disease is cellular-mediated autoimmune destruction of the pancreatic beta-cells.

The triggers for the autoimmune attack are not fully understood, but it is now widely accepted that both environmental and genetic factors contribute to it.

The strongest gene for type one diabetes mellitus, is located in the major histocompatibility complex Class II region on chromosome 6, at staining region 6p21.

Environmental factors can influence expression of type 1 diabetes and this can be suggested by the identical twins, when one twin has type 1 diabetes, the other twin only has it 30%-50% of the time.

It has been reported that only 10% of those who are genetically predisposed to type one diabetes actually develop the disease; however, that percentage appears to be changing and environmental factors may play an increasingly important role in determining risk.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with disease onset under the age of one year diagnosed according to American Diabetes Association criteria 2016 which include:
* Fasting plasma glucose level at or above 7.0 mmol/L (126 mg/dl).
* Plasma glucose at or above 11.1 mmol/L (200 mg/dl) two hours after a 1.75 gm/kg oral glucose load as in a glucose tolerance test.
* Symptoms of hyperglycemia and random plasma glucose at or above 11.1 mmol/L 200 mg/dl).
* Hemoglobin A1C at or above 48 mmol/mol.

Exclusion Criteria:

* Diabetic children with the disease onset above the age of one year.
* Infants with transient hyperglycemia.

Ages: 2 Months to 1 Year | Sex: All
Age Groups: Child
Study Population: Sixty diabetic patient diagnosed under the age of one year will be subjected for anti-insulin and anti-islets auto-antibodies who are negative for these test will be subjected to do genetic study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate possible risk factors among diabetic infants | within six months
  Questionnaire to evaluate possible risk factors among diabetic infants

SECONDARY OUTCOMES:
Detection of gene mutation responsible for infantile diabetes through gene sequencing | within six months
  Gene sequencing for detection of mutation in KCJN11 gene encoding the Kir6.2 subunit of adenosine tri-phosphate sensitive potassium channel.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No